CLINICAL TRIAL: NCT07322120
Title: Investigation of the Effect of Light Fasting Diet Combined With Magnesium Supplementation on Lipid Profile, Lipid Peroxidation, and C-Reactive Protein (CRP) Levels in Women With Polycystic Ovary Syndrome (PCOS).
Brief Title: Light Fasting Diet and Magnesium in Polycystic Ovary Syndrome (PCOS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Behnood Abbasi (Other)
Responsible Party: Sponsor-Investigator, Behnood Abbasi, Faculty member, Science & Research Islamic Azad University Branch Khozestan
Organization: Science & Research Islamic Azad University Branch Khozestan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.IAU.SRB.REC.1404.308
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Light Fasting; Magnesium; Lipid Profile; Lipid Peroxidation; C-Reactive Protein
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two parallel groups. Both groups follow a Light Fasting diet, but the intervention group receives magnesium supplementation, while the control group receives a placebo. The intervention lasts for 2 months, and primary outcomes include lipid profile, lipid peroxidation, and C-reactive protein (CRP) levels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a triple-blind study. Participants, investigators, and outcomes assessors are blinded to group allocation. Only the study coordinator has access to group assignments for safety purposes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light fasting and Magnesium Supplementation (Experimental): Participants follow a Light Fasting diet during the first month, designed with gradual caloric restriction and intermittent fasting days, followed by a maintenance diet tailored to individual needs during the second month. They receive magnesium supplementation (500 mg/day in two doses of 250 mg), for the full 2-month intervention.
  Interventions: Behavioral: Light fasting; Dietary Supplement: Magnesium supplementation
- Light fasting and Placebo (Placebo Comparator): Participants follow the same Light Fasting and maintenance diet schedule as the intervention group and receive a placebo supplement identical in appearance to the magnesium tablets, taken twice daily, for the full 2-month intervention.
  Interventions: Behavioral: Light fasting; Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Light fasting — Participants follow a Light Fasting diet during the first month, designed with gradual caloric restriction and intermittent fasting days, followed by a maintenance diet tailored to individual needs during the second month.
  Arms: Light fasting and Magnesium Supplementation
Dietary Supplement: Magnesium supplementation — Participants receive magnesium supplementation (500 mg/day in two doses of 250 mg), for the full 2-month intervention.
  Arms: Light fasting and Magnesium Supplementation
Behavioral: Light fasting — Participants follow a Light Fasting diet during the first month, designed with gradual caloric restriction and intermittent fasting days, followed by a maintenance diet tailored to individual needs during the second month.
  Arms: Light fasting and Placebo
Dietary Supplement: Placebo — Participants receive a placebo supplement identical in appearance to the magnesium tablets, taken twice daily, for the full 2-month intervention.
  Arms: Light fasting and Placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine disorders in women of reproductive age, which is associated with hormonal imbalances, dyslipidemia, chronic inflammation, and increased oxidative stress, and can increase the risk of cardiovascular and metabolic diseases. Evidence suggests that nutritional interventions play an important role in improving metabolic outcomes in these patients.

This study is a randomized, triple-blind, controlled clinical trial designed to investigate the effect of a light fasting diet combined with magnesium supplementation on lipid profile, lipid peroxidation (malondialdehyde), and C-reactive protein (CRP) levels in women with PCOS. In this study, 46 eligible women were randomly divided into two groups receiving a light fasting diet with magnesium supplementation or placebo, and changes in biochemical and anthropometric indices were evaluated before and after 8 weeks of intervention.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine and metabolic disorders in women of reproductive age, with a significant prevalence worldwide and in the Iranian female population. This syndrome is characterized by a set of hormonal and metabolic abnormalities, including hyperandrogenism, impaired ovulation, dyslipidemia, insulin resistance, mild chronic inflammation, and increased oxidative stress. Evidence suggests that women with Polycystic ovary syndrome (PCOS) have higher levels of inflammatory markers such as C-reactive protein (CRP) and lipid peroxidation indices such as malondialdehyde (MDA), and as a result, are at higher risk for cardiovascular and metabolic diseases. Currently, lifestyle modification including nutritional interventions and physical activity is recommended as the first line of treatment for Polycystic ovary syndrome (PCOS). Meanwhile, intermittent fasting-based diets, especially light fasting, have been proposed as a novel and sustainable approach that can improve lipid metabolism, reduce inflammation, and modulate oxidative stress without severe calorie restriction. On the other hand, magnesium, as an essential micronutrient, plays an important role in regulating glucose and lipid metabolism, increasing insulin sensitivity, reducing inflammation, and inhibiting oxidative processes. However, the evidence regarding the simultaneous effect of light fasting and magnesium supplementation on inflammatory markers and oxidative stress in women with Polycystic ovary syndrome (PCOS) is limited.

The present study is a randomized, triple-blind, controlled clinical trial designed to investigate the effect of light fasting combined with magnesium supplementation on lipid profile, lipid peroxidation, and C-reactive protein (CRP) levels in women with Polycystic ovary syndrome (PCOS). The study population includes women aged 19 to 65 years with Polycystic ovary syndrome (PCOS) with a body mass index equal to or higher than 25 kg/m2, diagnosed by a specialist based on the Rotterdam criteria. After obtaining informed consent, participants will be randomly divided into two groups. The intervention group will receive a light fasting diet with magnesium supplementation (500 mg/day in two doses of 250 mg), while the control group will receive the same light fasting diet with placebo. The nutritional intervention consists of a four-week cyclical program of light fasting designed to gradually adapt the body, and in the second month of the study, a diet with energy intake proportional to daily needs will be implemented to assess the sustainability of metabolic effects.

At the beginning of the study and after the end of the intervention period (8 weeks), anthropometric indicators including weight, Body mass index (BMI), and waist circumference will be measured. Physical activity was also assessed using the standard short-International physical activity questionnaire (IPAQ) and dietary intake was assessed using a three-day 24-hour food recall. Blood samples were collected after 12 to 14 hours of fasting and biochemical markers including total cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides, malondialdehyde (MDA), C-reactive protein (CRP), and luteinizing hormone (LH) and follicle-stimulating hormone (FSH) were measured using standard laboratory methods.

ELIGIBILITY:
Inclusion Criteria:

1. People between the ages of 19 and 65
2. People with a body mass index (BMI) ≤ 25
3. Diagnosis of polycystic ovary syndrome by a specialist based on the Rotterdam criteria

Exclusion Criteria:

1. Failure of the participant to cooperate during the study
2. Use of drug therapy that affects carbohydrate or fat metabolism (including oral contraceptives, insulin sensitizers, antiepileptic drugs, antipsychotics, statins, and fish oil) within the past 6 months.
3. Planning for pregnancy, pregnant, or breastfeeding
4. In the perimenopausal stage
5. Low blood pressure
6. Presence of other diseases (such as congenital adrenal hyperplasia, Cushing's syndrome, androgen-secreting tumors, hyperprolactinemia, diabetes, thyroid disease, severe cardiovascular, gastrointestinal, renal, and hepatic diseases)
7. Performing high-intensity exercise

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of total cholesterol | Baseline and 8 weeks after
  Serum TC (total cholesterol) concentration (mg/dl)

SECONDARY OUTCOMES:
Change from baseline of Triglyceride | Baseline and 8 weeks after
  Serum TG (triacylglycerol) concentration (mg/dl)
Change from baseline of low density lipoprotein cholesterol (LDL-Cholesterol) | Baseline and 8 weeks after
  Serum LDL concentration (mg/dl)
Change from baseline of high density lipoprotein cholesterol (HDL-Cholesterol) | Baseline and 8 weeks after
  Serum HDL concentration (mg/dl)
Change from baseline of Lipid Peroxidation | Baseline and 8 weeks after
  Changes in serum levels of lipid peroxidation markers (e.g., MDA)
CRP | Baseline and 8 weeks after
  Changes in serum levels of C-reactive protein (CRP)

IPD SHARING:
Plan to Share IPD: No